CLINICAL TRIAL: NCT00546065
Title: APE-Study: Tumor-free Survival After Ablation of Barrett's Mucosa Plus Esomeprazole vs. Surveillance Without Ablation in Patients Cured From Barrett's Cancer Combined With Randomization of Esomeprazole vs Placebo for Symptomatic Reflux Control After Successful Ablation of Barrett's Mucosa
Brief Title: APE-Study: Ablation of Barrett's Mucosa vs. Surveillance Without Ablation in Patients Cured From Barrett's Cancer Combined With Randomization of Esomeprazole vs. Placebo for Symptomatic Reflux Control After Successful Barrett's Ablation
Acronym: APE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intermediate results have shown a significant difference in the outcome of ablation and non-ablation patients. Therefore, the study was stopped.
Sponsor: HSK Wiesbaden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D9612L00088
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's esophagus; ablation; esomeprazole; Barrett's cancer; Ablation of Barrett's esophagus; Surveillance of Barrett's esophagus after endoscopic resection of Barrett's cancer; Recurrence of Barrett's cancer
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ablation of Barretts with concomitant esomeprazole therapy (Other): comparison of recurrence-free survival
  Interventions: Drug: esomeprazole treatment
- non ablation (No Intervention): non ablation only surveillance
  Interventions: Drug: esomeprazole treatment

INTERVENTIONS:
Drug: esomeprazole treatment — concomitant esomeprazole treatment

SUMMARY:
This is a prospective, randomized, controlled, double-blinded, multi-center trial in a parallel-group design. Aim of the study is the evaluation of tumor-free survival after ablation (by APC, argon plasma coagulation) of Barrett's mucosa plus esomeprazole versus surveillance without ablation in patients cured from Barrett's cancer combined with randomization of esomeprazole vs placebo for symptomatic reflux control after successful ablation of Barrett's mucosa .

There are two hypotheses: (1) Consecutive thermal ablation of metaplastic, non-neoplastic long segments of Barrett's esophagus (>2cm)plus esomeprazole after successful endoscopic therapy of mucosal cancer by means of ER will decrease the incidence of secondary cancer (local recurrence and metachronous cancer) by a minimum of 50% compared to acid suppression alone without ablation within a 5-years follow-up (primary endpoint). (2) After successful ablation of Barrett's esophagus patients need ongoing acid suppression therapy for medical control of their underlying reflux disease (secondary aim of the study).

Duration of the study:

Patient recruitment period: 3 years. Follow-up period: 5 years. Total duration: 8 years. The study is already in the recruitment period.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopically and histologically complete remission of mucosal Barrett's cancer (endoscopic resection with or without thermal ablation of resection margins)
* Initial length of Barrett's segment before cancer therapy > 3 cm (initially long-segment Barrett's esophagus)
* Barrett's length after endoscopic therapy of Barrett's cancer > 2 cm
* Informed consent of the patient

Exclusion Criteria:

* Attempted ablation therapy before the trial
* Treatment duration of early Barrett's cancer > 12 months
* Duration between achievement of complete remission and attempted inclusion into the study > 24 months
* The Barrett's cancer treated has already been a secondary lesion of earlier Barrett's cancer
* Inadequate healing of endoscopic resection (ER) ulcers
* No residual Barrett's mucosa observed after pretreatment with ER
* No PPI compliance
* Relevant comorbidity (e.g., malignancy)
* Pregnancy
* Age below 18 years
* Patient not able to understand study characteristics
* No written informed consent available
* Allergy against esomeprazole or intolerance of medication ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
recurrence-free survival | 3 years
  recurrence-free survival during 3 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ell, MD PhD, Principal Investigator — HSK Wiesbaden
Locations (1):
- HSK Wiesbaden, Wiesbaden, Hesse, Germany